CLINICAL TRIAL: NCT06185491
Title: Assessment of HGI (Hemoglobin Glycation Index) Variability Over Time in Patients Living With Diabetes Using Continuous Glucose Monitoring
Brief Title: Assessment of HGI (Hemoglobin Glycation Index) Variability Over Time in Patients Living With Diabetes Using Continuous Glucose Monitoring ( GAP OUEST )
Acronym: GAP OUEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC22_0502
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HGI (Experimental): Data collection from glucose monitoring systems. Dosage of glycated hemoglobin and glycated albumin
  Interventions: Other: HGI

INTERVENTIONS:
Other: HGI — Data collection from glucose monitoring systems and dosage of glycated hemoglobin and glycated albumin measured 3 times at 6-month intervals (+/- 3 months)

SUMMARY:
The goal of this clinical trial is to learn about the variability of HGI (Hemoglobin Glycation Index) over time in patients living with diabetes using a continuous glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Major (adult subject over 18), with no upper age limit
* Enrolled in a social security scheme or beneficiary of such a scheme
* Agreement to participate (informed, written consent)
* Established diabetes (regardless the type of diabetes), known for at least 6 months at inclusion
* Regular user of a glucose monitoring system for at least 3 months.

Non inclusion Criteria:

* Known hemoglobinopathy
* Inadequate use of the flash glucose monitoring system with a capture rate of less than 70% of interstitial glucose measurements, during the 3 months preceding the inclusion visit.
* Stage 5 renal insufficiency (CKD-EPI less than 15 mL/min/1.73 m2)
* Pregnant or breast-feeding
* Major under guardianship, curatorship or safeguard of justice
* Any situation assessed by the investigator as potentially prejudicial to the participant's health as a result of participation in the study

Exclusion criteria:

* Treatment with corticosteroids in the 3 months preceding the visit
* Unusual acute situation (infection, very unusual physical activity, etc.) deemed significant by the investigator
* Pregnancy started

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Coefficient of variation of individual HGI distribution | 12 months
  calculated from 3 HGI values, measured 6 months apart, HGI = HbA1C measured in laboratory - HbA1C estimated

SECONDARY OUTCOMES:
Coefficient of variation of the individual distribution of the albumin glycation index | 12 months
  Albumin glycation index = glycated albumin measured in laboratory - glycated albumine estimated
Glycation gap, determined from comparison between HbA1C measured and HbA1C derived from glycated albumin | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hélène AUFFRET, Principal Investigator — Nantes University Hospital
Locations (10):
- France (10):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CH de La Rochelle, La Rochelle
  - CH du Mans, Le Mans
  - CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - Hôpital NOVO, Pontoise
  - CHU de Rennes, Rennes
  - CHU de Toulouse, Toulouse